CLINICAL TRIAL: NCT06604312
Title: The Immediate Effect of Sacroiliac Joint Manipulation on Postural Balance, Range of Motion and Muscle Strength in Standing Workers
Brief Title: The Immediate Effect of Sacroiliac Joint Manipulation in Standing Workers
Acronym: IESJMSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SEFA HAKTAN HATIK (Other)
Responsible Party: Sponsor-Investigator, SEFA HAKTAN HATIK, Assistant Professor, Sinop University
Organization: Sinop University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CMT0005
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Neuromuscular Subluxation of Joint; Physical Therapy
Keywords: Chiropractic; Sacroiliac joint; Postural balance; Muscle strength

STUDY DESIGN:
Intervention Model Description: Forty volunteers participated in the study and these participants were divided into sacroiliac joint manipulation group (n=20) and control group (n=20). The sacroiliac joint manipulation was performed in the lateral decubitus position and the control group did not underwent any manipulation. Assessment methods were performed immediately after the manipulation. The frequency and percentage values for categorical variables and the mean, standard deviation, and median values for numerical data were displayed, respectively. Since there were less than thirty data points in each group, nonparametric tests were used to examine the data. The Mann-Whitney U test was used to compare the data between the two groups, and the Wilcoxon sign test was utilized to examine the difference between the two measures for each group. Measurement time differences were recorded, and the Mann-Whitney Test was used to compare the groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacroiliac Joint Manipulation Group (Experimental): Sacroiliac joint manipulation was performed in lateral decubitis position.
  Interventions: Other: Sacroiliac Joint Manipulation
- Control Group (No Intervention): The control group did not undergo any treatment.

INTERVENTIONS:
Other: Sacroiliac Joint Manipulation — Sacroiliac manipulation was performed using manual treatment method by lying patients on their sides. First, the patient was positioned firmly on the edge of the examination table, while the restricted sacroiliac joint remains on the upper side. Then, the physician's hand was positioned on the patient's hip, and the flexion was made on the lumbar spine with the movement from the hip to the upper thigh, and the impulse given by the HVLA technique was applied in the anteroinferior direction to the iliac crest and trochanter major.
  Arms: Sacroiliac Joint Manipulation Group

SUMMARY:
The aim of this study was to determine whether sacroiliac joint manipulation has a positive effect on muscle strength, balance and range of motion in standing workers.

DETAILED DESCRIPTION:
The study included 40 participants who were previously informed about the study, met the inclusion criteria and signed the consent form. Participants were randomly divided into two groups as sacroiliac joint manipulation group (n=20) and control group (n=20). Hip and lumbar range of motion was assessed with a goniometer, postural control and balance with Biodex, and quadriceps femoris and hamstring muscle strength with MicroFet®2. The sacroiliac joint manipulation group underwent sacroiliac joint manipulation and the control group did not undergo any procedure. The effect of the manipulation was measured immediately after the manipulation and the significance level was accepted as p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* Having signed the voluntary consent form
* Being between the ages of 18-50
* Working standing for at least 3 hours a day
* Working standing for at least 6 months
* Suffering from low back pain in the last 6 months.

Exclusion Criteria:

* Having diseases that may cause balance problems
* Having a history of trauma in the last 6 months
* Pregnancy or suspicion of pregnancy
* Contraindications to chiropractic treatment (such as tumor, rheumatological condition, fracture, dislocation, metastasis and aneurysm)
* Feeling pain in the pelvis and sacroiliac joint,

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Biodex Balance System | It was performed immediately after the manipulation. In the control group, the first measurement was performed and the second measurement was repeated after waiting for 15 minutes.
  Biodex Balance System (Biodex, Inc, Shirley, New York) (BDS) device was used to measure postural balance. It can extract anterior-posterior stability index (APSI), mediolateral stability index (MLSI) and overall stability index (OSI) for the measurement of standing posture control. Lower oscillation scores indicate better postural stability (Sung and Kim, 2018). The bipedal balance tests were performed with eyes open and closed and the volunteers were measured with their hands at their sides. The tests were performed for 30 seconds.
Muscle Strength | It was performed immediately after the manipulation. In the control group, the first measurement was performed and the second measurement was repeated after waiting for 15 minutes.
  Muscle strength measurements were performed with microFET ®2, a digital handheld dynamometer. The measurement is based on the compression principle and has high reliability and measurement accuracy. The results were recorded in kilograms of force (kgf) and measurements were taken from the quadriceps femoris and hamstring muscles.
Range of Motion | It was performed immediately after the manipulation. In the control group, the first measurement was performed and the second measurement was repeated after waiting for 15 minutes.
  Range of motion (ROM) measurements were performed with a universal goniometer. Degree was used as the unit of measurement. Flexion, extension, internal rotation, external rotation, abduction and adduction angles were measured bilaterally for the hip joint. Flexion, extension and lateral flexion (left-right) were measured in the lumbar region. For these values, the values determined by the American Association of Orthopedic Surgeons were taken as a basis, recorded during the measurement and proceeded in order.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinop University, Sinop, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes